CLINICAL TRIAL: NCT03425539
Title: A Multicenter, dOuble-blind, ranDomized, Placebo-controlled, Parallel-group Study to Determine the effIcacy and Safety of Lucerastat Oral Monotherapy in Adult Subjects With FabrY Disease
Brief Title: Efficacy and Safety of Lucerastat Oral Monotherapy in Adult Subjects With Fabry Disease
Acronym: MODIFY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-069A301
Record Dates: First submitted 2018-01-16; First posted 2018-02-07 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — migalastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lucerastat (Experimental)
  Interventions: Drug: Lucerastat
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lucerastat — Hard gelatin capsules containing 250 mg of lucerastat and inactive excipients; 1000 mg (4 capsules) twice daily (b.i.d.); dose adjusted for renal function.
  Arms: Lucerastat
Drug: Placebo — Placebo capsules are identical in appearance to the lucerastat capsules, and contain inactive excipients; 4 capsules b.i.d.; dose adjusted for renal function.
  Arms: Placebo

SUMMARY:
This study aimed to determine the efficacy and safety of lucerastat oral monotherapy in adult subjects with Fabry disease.

DETAILED DESCRIPTION:
The primary objective of this prospective, multicenter, double-blind, randomized, placebo-controlled, parallel group, Phase 3 study is to determine the effect of oral lucerastat monotherapy on neuropathic pain in subjects with Fabry disease (FD) through daily collection of patient-reported outcomes with an electronic diary.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated ICF prior to any study-mandated procedure;
2. Male or female adult subjects;
3. FD diagnosis confirmed with local genetic test results;
4. Fabry-associated neuropathic pain, as defined by the subject, in the last 3 months prior to screening;
5. Enzyme replacement therapy (ERT) status:

   1. Subject never treated with ERT; or
   2. Subject has not received ERT for at least 6 months prior to screening; or
   3. Subject treated with ERT since at least 12 months at the time of the screening visit, and agreeing to stop ERT for approximately 8 months.
6. A woman of childbearing potential is eligible only under certain conditions, e.g. taking contraceptive measures.
7. Subjects with moderate or severe neuropathic pain during the screening period.

Exclusion Criteria:

1. Pregnant, planning to be become pregnant, or lactating subject.
2. Severe renal insufficiency (eGFR < 30 mL/min/1.73 m2) at screening.
3. Subject on regular dialysis for the treatment of chronic kidney disease.
4. Known and documented transient ischemic attack, stroke, unstable angina, or myocardial infarction within 6 months prior to screening.
5. Clinically significant unstable cardiac disease (e.g. uncontrolled symptomatic arrhythmia, congestive heart failure NYHA class III or IV).
6. Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (49):
- United States (17):
  - University of Alabama at Birmingham - Nephrology Research Clinic, Birmingham, Alabama
  - University of California Irvine, Irvine, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of Florida College of Medicine - Division of Nephrology, Hypertension & Renal Transplantation, Gainesville, Florida
  - Emory University School of Medicine; Department of Human Genetics, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Stead Family Children's Hospital - Division of Medical Genetics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Infusion Associates, Grand Rapids, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh (UPMC), Pittsburgh, Pennsylvania
  - Greenwood Genetic Center, Greenville, South Carolina
  - Research Baylor Institute of Metabolic Disease, Dallas, Texas
  - University of Utah - Division of Medical Genetics, Salt Lake City, Utah
  - Lysosomal and Rare Disorders Research and Treatment Center, Fairfax, Virginia
- Australia (2):
  - Royal Melbourne Hospital - Department of Nephrology, Parkville
  - Royal Perth Hospital, Department of Nephrology, Perth
- Allgemeines Krankenhaus der Stadt Wien - Universitätsklinik für Innere Medizin III - Klinische Abteilung für Nephrologie und Dialyse, Vienna, Austria
- Belgium (2):
  - University Hospital Ghent, Ghent
  - University Hospital Leuven, Leuven
- Canada (6):
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - M.A.G.I.C Clinic Ltd, Calgary
  - Queen Elizabeth II Health Sciences Center - Halifax Infirmary - Division of Nephrology, Halifax
  - Research Center, Hôpital Du Sacré-Coeur de Montréal, Montreal
  - Vancouver Hospital & Health Sciences - Vancouver General Hospital, Vancouver
  - Health Sciences Center Winnipeg, Winnipeg
- Germany (4):
  - Charite Campus Virchow-Klinikum - Nephrologie und Internistische Intensivmedizin, Berlin
  - SphinCS GmbH, Höchheim
  - Fachinternistische Gemeinschaftspraxis Markgräferland, Mühlheim
  - Medizinische Klinik und Poliklinik I der Universität - Schwerpunkt Nephrologie, Würzburg
- Hosp Alma Mater Studiorum, Dublin, Ireland
- Italy (2):
  - ASST Monza, Hospital San Gerardo, Nephrology, Monza
  - University of Naples Federico II (Nephrology), Naples
- Hospital Academisch Medisch Centrum - Department of Internal Medicine Div. Endrocrinology and Metabolism, Amsterdam, Netherlands
- Haukeland University Hospital Helse Bergen HF, Bergen, Norway
- Poland (3):
  - University Hospital in Cracow - Dep. of of Allergies and Immunology, Krakow
  - Cardinal Wyszynski Institute of Cardiology, Warsaw
  - Department of Pediatric Nutrition and Metabolic Diseases; The Children's Memorial Health Institute, Warsaw
- Spain (4):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Universitari de Bellvitge; Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Ramon y Cajal. Servicio de Medicina Interna, Madrid
  - Hospital Quironsalud Zaragoza, Zaragoza
- Universität Zürich Psychiatrische Universitätsklinik, Zurich, Switzerland
- United Kingdom (4):
  - University Hospital Birmingham NHS Foundation Trust - Center for Rare Diseases, Birmingham
  - The Royal Free Hospital, Department of Haematology Royal Free London NHS Foundation Trust, London
  - National Hospital for Neurology and Neurosurgery, London
  - Salford Royal (Hope) Hospital, Salford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 49 sites in 14 countries, including North America (USA, CAN), Europe (Austria, Belgium, Germany, Ireland, Italy, Netherlands, Norway, Poland, Spain, Switzerland, UK), and Australia.
Groups:
- Lucerastat: Lucerastat (ACT-434964) was provided as hard-gelatin capsules containing 250 mg of lucerastat.
  Capsules were administered orally twice daily (b.i.d.) to provide a lucerastat dose of 250, 500, 750, or 1000 mg b.i.d. based on the subject's estimated glomerular filtration rate (eGFR).
- Placebo: Matching placebo capsules were administered orally b.i.d., with the number of capsules administered based on the subject's eGFR.
Period: Overall Study
Arm/Group | Lucerastat | Placebo
Started | 80 | 38
Treated | 80 | 37
Completed | 75 | 34
Not Completed | 5 | 4
Not completed — Randomized but not treated | 0 | 1
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lucerastat: Lucerastat (ACT-434964) was provided as hard-gelatin capsules containing 250 mg of lucerastat.
  Capsules were administered orally b.i.d. to provide a lucerastat dose of 250, 500, 750, or 1000 mg b.i.d. based on the subject's eGFR.
- Total: Total of all reporting groups
Arm/Group | Lucerastat | Placebo | Total
Number analyzed (Participants) | 80 | 38 | 118
Age, Continuous [Median (Full Range); unit: years] | 38 [18 to 74] | 39 [18 to 65] | 39 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 20 | 63
  Male | 37 | 18 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 76 | 37 | 113
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 26 | 6 | 32
  United Kingdom | 8 | 3 | 11
  Switzerland | 0 | 1 | 1
  Spain | 7 | 6 | 13
  Canada | 10 | 5 | 15
  Netherlands | 1 | 2 | 3
  Austria | 0 | 1 | 1
  Belgium | 3 | 1 | 4
  Norway | 1 | 1 | 2
  Poland | 9 | 4 | 13
  Australia | 5 | 4 | 9
  Germany | 10 | 4 | 14
Neuropathic pain monthly score at baseline [Mean (Standard Deviation); unit: units on a scale] — Neuropathic pain on the modified Brief Pain Inventory-Short Form 3 (modified BPI-SF3): subjects rated their neuropathic pain intensity ("neuropathic pain at its worst in the last 24 hours") on an 11-point scale, from 0 (no neuropathic pain) to 10 (worst imaginable neuropathic pain).
  units on a scale | 6.26 (1.54) | 6.11 (1.39) | 6.21 (1.49)

OUTCOME MEASURES:

1. Primary Outcome: Neuropathic Pain Monthly Score: Change From Baseline to Month 6
Description: Neuropathic pain on the modified BPI-SF3: subjects rated their neuropathic pain intensity ("neuropathic pain at its worst in the last 24 hours") on an 11-point scale, from 0 (no neuropathic pain) to 10 (worst imaginable neuropathic pain).
Time Frame: From baseline to Month 6 (duration: 6 months)
Population: The analysis included all subjects who were randomized and took at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lucerastat | Placebo
Number analyzed (Participants) | 80 | 37
score on a scale | -1.64 [-2.11 to -1.16] | -2.05 [-2.73 to -1.37]
Statistical Analysis 1: Comparison: Lucerastat vs Placebo; Test type: Other — An ANCOVA was applied to the change from baseline to Month 6 including the baseline value, the two stratification factors (sex and enzyme replacement therapy (ERT) treatment status), and the treatment group; p = 0.3189, ANCOVA; LS Mean difference vs. placebo = 0.42, 95% CI 2-sided [-0.4 to 1.23]

2. Secondary Outcome: Plasma Globotriaosylceramide (Gb3; in ng/ml): Change From Baseline to Month 6
Time Frame: From baseline to Month 6 (duration: 6 months)
Population: The analysis included all subjects who were randomized and took at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Lucerastat | Placebo
Number analyzed (Participants) | 80 | 37
ng/ml | -672.68 [-798.91 to -546.46] | 200.84 [14.29 to 387.40]
Statistical Analysis 1: Comparison: Lucerastat vs Placebo; Test type: Other — An ANCOVA was applied to the change from baseline to Month 6 including the baseline value, the two stratification factors (sex and ERT treatment status), and the treatment group; p < 0.0001, ANCOVA; LS Mean difference vs. placebo = -873.53, 95% CI 2-sided [-1097.53 to -649.53]

3. Secondary Outcome: Abdominal Pain Monthly Score: Change From Baseline to Month 6
Description: Abdominal pain on the 11-point Numerical Rating Scale (NRS-11): subjects rated their abdominal pain intensity ("abdominal pain at its worst in the last 24 hours") on an 11-point scale, from 0 (no pain) to 10 (worst imaginable pain).
Time Frame: From baseline to Month 6 (duration: 6 months)
Population: The analysis included randomized and treated subjects with gastrointestinal symptoms at baseline (diarrhea on at least 8 days and/or moderate or severe abdominal pain in the 4 weeks prior to randomization).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lucerastat | Placebo
Number analyzed (Participants) | 61 | 29
score on a scale | -1.37 [-1.86 to -0.87] | -1.68 [-2.38 to -0.98]
Statistical Analysis 1: Comparison: Lucerastat vs Placebo; Test type: Other — An ANCOVA was applied to the change from baseline to Month 6 including the terms value, the two stratification factors (sex and ERT treatment status), and the treatment group; p = 0.4676, ANCOVA; LS Mean difference vs. placebo = 0.31, 95% CI 2-sided [-0.53 to 1.16]

4. Secondary Outcome: Number of Days With Diarrhea: Change From Baseline to Month 6
Description: A subject was considered to have diarrhea on a specific day if at least one stool of a Bristol Stool Scale (BSS) consistency Type 6 or 7 was reported. The number of days with diarrhea at baseline and Month 6 was the number of days with diarrhea over the 4 weeks prior to the randomization visit or the Month 6 visit, respectively, adjusted for the number of days with data available.
Time Frame: From baseline to Month 6 (duration: 6 months)
Population: The analysis included randomized and treated subjects with gastrointestinal symptoms at baseline (diarrhea on at least 8 days and/or moderate or severe abdominal pain in the 4 weeks prior to randomization) and a non-missing change from baseline to Month 6 value.
Measure: Mean (Standard Deviation); unit: Number of days within 4 weeks
Arm/Group | Lucerastat | Placebo
Number analyzed (Participants) | 48 | 25
Number of days within 4 weeks | -3.45 (4.96) | -3.95 (9.29)
Statistical Analysis 1: Comparison: Lucerastat vs Placebo; The p-value was derived from a rank ANCOVA adjusted for the baseline value and stratified by sex and ERT treatment status; Test type: Other; p = 0.8986, ANCOVA; Win ratio = 1.00, 95% CI 2-sided [0.57 to 1.89]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events from the 6-month treatment period are reported. Adverse events were considered treatment-emergent if the onset date was between the first intake of study treatment up to 30 days after the end of study treatment.
Description: Adverse events for all subjects in the lucerastat arm are reported together, regardless of dose. This is due to the study treatment dosing scheme, where each subject's dose of study treatment was based on their individual eGFR.
Arm/Group | Lucerastat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/37
Serious Adverse Events (participants affected / at risk) | 5/80 | 1/37
Other Adverse Events (participants affected / at risk) | 46/80 | 21/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lucerastat (N=80) | Placebo (N=37)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Septic encephalopathy (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lucerastat (N=80) | Placebo (N=37)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 1 (1)
Flatulence (Gastrointestinal disorders) | 7 (7) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (13) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7) | 0 (0)
Fatigue (General disorders) | 3 (3) | 6 (7)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 8 (10) | 5 (5)
Vaccination complication (Injury, poisoning and procedural complications) | 5 (10) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (3)
Headache (Nervous system disorders) | 9 (11) | 4 (4)
Neuralgia (Nervous system disorders) | 6 (6) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to the sponsor for review at least 30 days prior to submission for publication or presentation at a congress. Upon review, the sponsor may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator should permit publication during such a review period.

DOCUMENTS (2):
  • Study Protocol (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT03425539/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT03425539/SAP_001.pdf